CLINICAL TRIAL: NCT05929014
Title: The Effect of Different Intensities of Bilateral-transcranial Direct Current Stimulation (tDCS) on Cortical Activity and Motor Learning in Healthy Individuals
Brief Title: Effects of Different Intensities of Bilateral-transcranial Direct Current Stimulation in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MU-CIRB 2023/016.1601
Record Dates: First submitted 2023-06-25; First posted 2023-07-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: tDCS; Cortical activity; Healthy; Motor learning; Brain symmetry index

STUDY DESIGN:
Intervention Model Description: The participants who will participate in the study will be randomly received 1 mA or 1.5 mA or 2 mA or sham with the washout period for at least 2 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active bilateral-tDCS (Active Comparator): Participants will be received different intensities which are 1 mA, 1.5 mA and 2 mA for 20 minutes during performed serial reaction time task. The tDCS will be set with bilateral montage which applied anodal electrode over left hemisphere and cathodal electrode over right hemisphere.
  Interventions: Device: Bilateral-Transcranial direct current stimulation (bilateral-tDCS)
- Sham bilateral-tDCS (Sham Comparator): Participants will be received sham of bilateral tDCS during performed serial reaction time task.
  Interventions: Device: Sham bilateral-tDCS

INTERVENTIONS:
Device: Bilateral-Transcranial direct current stimulation (bilateral-tDCS) — The tDCS is non-invasive brain stimulation technique applied over the participant's scalp using a reference to the International 10-20 electrode Placement System for EEG electrode placement. The cathodal and anodal electrodes will be applied over the right and left primary motor areas, respectively.
  Other Names: MINDD STIM; Ybrain Inc., Korea
  Arms: Active bilateral-tDCS
Device: Sham bilateral-tDCS — Sham bilateral-tDCS
  Arms: Sham bilateral-tDCS

SUMMARY:
This study will investigate the effects of 1 mA, 1.5 mA, and 2 mA of bilateral- tDCS on cortical activity and motor learning in healthy individuals

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is one of the non-invasive brain stimulation (NIBS) techniques. It delivers weak direct current through the scalp via two electrodes. tDCS has been shown to modulate cortical excitability in polarity-specific effects; anodal increases cortical excitability, while cathodal decreases it. tDCS can be applied in two distinct montages: unilateral (an active electrode is applied over the cerebral cortex, while a reference electrode is applied over the contralateral orbit) and bilateral-tDCS (applying two electrodes simultaneously over both cerebral hemispheres). Many tDCS studies have been used as an add-on therapy in stroke patients which aimed to enhance motor re-learning after stroke. Anodal tDCS has been used to enhance cortical excitability in the lesioned hemisphere while cathodal tDCS is used to decrease it in the non-lesioned hemisphere and thus to rebalance the interhemispheric inhibition (IHI). However, there were recent studies reporting the reverse effect of cathodal-tDCS on cortical excitability at high doses. However, the effects of bilateral-tDCS among different doses on cortical excitability and on motor performance are still controversial.

The present study will be investigated the effects of different intensities of bilateral-tDCS on cortical activity and functional outcomes in healthy individuals. A single session of different intensities of bilateral-tDCS (i.e., 1 mA, 1.5 mA, 2 mA vs. sham) will be combined with serial reaction time task (SRTT) in healthy individuals. Cortical activity (i.e., brain symmetry index (BSI)) will be measured as a primary outcome. The reaction time of serial reaction time task will be served as the secondary outcome. Cortical activity will be evaluated before and after the intervention, while reaction time will be evaluated before, during, and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-29 years old
* 2. Righ-hand dominant according to the Edinburgh handedness inventory
* 3. No injury to both upper and lower limb for the past 6 months

Exclusion Criteria:

* 1. Presence of any neurological disorders
* 2. Presence of metal implantation, intracranial shunt, cochlear implantation, or cardiac pacemakers
* 3. Presence of opened wound or infectious wound around scalp
* 4. History of epilepsy or any neurological antecedent or unstable condition which can lead to seizure
* 5. Body mass index (BMI) > 30 kg/m2
* 6. Received hormonal treatment and/or drugs that increase sleepiness and affect movement control
* 7. Ischemic heart disease and peripheral vascular ischemia
* 8. Last stage of kidney disease and liver disease

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-24 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Cortical activity | 5 minutes
  Acquired by electroencephalography (EEG)
The reaction time | 30 minutes
  Measured the reaction time from serial reaction time task

CONTACTS AND LOCATIONS:
Overall Officials: Wanalee Klomjai, PhD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Nakonpathom, Thailand

IPD SHARING:
Plan to Share IPD: No